CLINICAL TRIAL: NCT06964204
Title: The Effect of Kangaroo Care and Lullaby on Mother-Baby Physiological Parameters and Mother's State Anxiety Level in Premature Newborns: A Randomized Controlled Study
Brief Title: The Effect of Kangaroo Care and Lullaby on Mother-Baby Physiological Parameters and Mother's State Anxiety Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Edanur Tar Bolacali, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SU-2025-041
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: The Gestational Age of the Newborn is Between 28-37 Weeks; Stable Health Status of the Newborn; Mothers' Willingness to Participate in the Study
Keywords: Infant, Premature; Kangaroo-Mother Care Method; Lullabies; Physiological Parameters; Anxiety
MeSH Terms: conditions — Premature Birth; Anxiety Disorders | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: The sample of the study will be selected by "random sampling" method from mothers and their babies who are diagnosed and treated in the NICU of Osmaniye State Hospital and who meet the criteria for acceptance into the study. The sample size of the study was calculated as a total of 57 newborns in the G*Power 3.1.9.2. program with reference to a similar study in the literature (Arnon, 2014), which is parallel to our study. In the study, in order to reduce selection bias and control variables that may have an effect on the outcome parameters, the groups will be named as A and B and newborns will be randomly assigned to these groups. A: kangaroo care and B: kangaroo care+nurture or B: kangaroo care and A: kangaroo care+nurture will be determined by lottery. Before the study, mothers will be informed about both groups during the informed consent process and it will not be specified which group the newborns will be in.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo Care (Experimental): Kangaroo care will be applied to the babies in the 1st group and inclusion in the groups will be done by randomization.
  Interventions: Behavioral: Kangaroo Care
- Kangaroo Care + Lullaby (Experimental): In addition to kangaroo care, mothers will sing a lullaby to the babies in the 2nd group and inclusion in the groups will be done by randomization.
  Interventions: Behavioral: Kangaroo Care+lullabies

INTERVENTIONS:
Behavioral: Kangaroo Care — Kangaroo care practice will be carried out in 3 stages: "preparation, implementation and recording stage". Vital signs of the baby such as body temperature, heart rate, respiratory rate will be evaluated and necessary materials such as hats and covers will be prepared. In the implementation phase; the general condition of the baby will be checked, clothing and position will be adjusted, and then the baby will be transferred to the mother. After the baby is placed, his/her back will be covered with a blanket and the mother will be asked to support the baby's back with one hand and the hips with the other. When 60 minutes are completed, kangaroo care will be terminated. After the baby is placed, vital signs and general condition will be evaluated and all nursing observations will be recorded. For the babies in the other group, their mothers will sing lullabies along with kangaroo care and inclusion in the groups will be done by randomization.
  Arms: Kangaroo Care
Behavioral: Kangaroo Care+lullabies — For the babies in the other group, their mothers will sing lullabies along with kangaroo care and inclusion in the groups will be done by randomization.
  Arms: Kangaroo Care + Lullaby

SUMMARY:
This study was planned to investigate the effect of kangaroo care and lullaby on mother-baby physiologic parameters and mother's state anxiety level in premature newborns.

DETAILED DESCRIPTION:
Due to health problems, premature infants are subjected to many painful and uncomfortable interventions such as intubation and respiratory support, umbilical catheter, intravenous interventions, nasogastric catheter, sometimes gastrostomy, peritoneal dialysis, eye examinations and operations. The premature newborn may therefore be deprived of compassionate care that will provide comfort, such as sucking, cuddling, touching and eye contact, which are basic needs. The mother-infant relationship may be negatively affected because premature babies are different from what is imagined and have some health problems and are transferred to the intensive care unit. The birth of a premature baby, which is a crisis for the whole family, can cause intense anxiety and fear that the mother will lose her baby. The mother may avoid touching her baby for fear of harming her baby, and participating in the care of her baby can be very difficult and anxiety-provoking. Nurses working in the neonatal service and neonatal intensive care unit play a major role in ensuring mother-infant interaction in premature babies. It should enable the mother to share the same room (rooming-in), skin-to-skin contact (kangaroo care), eye-to-eye contact, hugging her baby, participating in the care of her baby and maintaining breastfeeding, which will increase the intimacy between mother and baby. Kangaroo care is a method in which newborns are placed on their mothers' chests, facing the mother, and skin-to-skin contact between mother and baby is ensured in order to ensure the early discharge of the baby from the hospital and to ensure that the baby starts to benefit from breast milk as soon as possible. Kangaroo care should be initiated as early as possible in the delivery room or neonatal intensive care unit to ensure thermal regulation, physiological stability, appropriate stimulation and to increase the rate of attachment and breastfeeding. It is known that the fetus recognizes the mother's voice from the 32nd week of gestation and in the postnatal period and responds with parameters such as increased pulse rate. It is argued that lullaby recital in neonatal intensive care has a relaxing effect on the newborn by masking environmental stressors and negative sounds. During kangaroo care, the baby's ear rests directly against the mother's breast, skin-to-skin contact and sounds are transferred to the baby through tissue and air, and the mother's voice is compared to the fetal auditory environment that the baby hears in the uterus, and it is thought that the positive effects on the mother and baby should be examined. This study was planned to examine the effect of kangaroo care and lullaby on the physiologic parameters of the mother and infant and the mother's state anxiety level in premature newborns. Thus, it is aimed to provide physiological stability in the infant and to increase mother-infant bonding by determining the effect of kangaroo care and lullaby, which are safe, inexpensive and easily applicable methods, on the vital signs of the mother and infant and the anxiety level of the mother.

ELIGIBILITY:
Inclusion Criteria:

* The gestational age of the newborn is between 28-37 weeks,
* Stable health status of the newborn,
* Mothers' willingness to participate in the study.

Exclusion Criteria:

* The gestational week of the newborn is below 28 weeks and above 37 weeks
* Unstable health status of the newborn,
* Hospitalization for at least 3 days,
* Parents were not willing to participate in the study.

Exclusion Criteria (during the research):

* Sudden need for resuscitation
* Sudden deterioration of the stabilization of health status

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
1. Mother and Newborn Introductory Information Form | First measurement - Before starting the study
  The form prepared by the researcher in line with the literature (Arnon et al., 2014) consists of a total of 22 questions about the mother and the infant. The questions questioning the characteristics of the mother in the form are "age, educational status, occupation, family type, presence of social security, economic status, disease status, number of pregnancies, whether the last pregnancy was planned, and when she breastfed her baby for the first time after birth". The questions about the infant consisted of "gender, gestational age, postnatal age, mode of delivery, 1st and 5th minute APGAR score, birth and weight, height, head circumference, hospitalization diagnosis and duration, and infant's diet". The form was sent to 5 academicians specialized in Pediatric Nursing and their expert opinions were obtained, and the information form was finalized in line with their suggestions.

SECONDARY OUTCOMES:
2. Mother Infant Physiologic Parameters Monitoring Form | Before and after the intervention for 3 days after starting the study
  The chart was created by the researcher to monitor the physiologic parameters of the newborn according to the type of intervention (kangaroo care - lullaby with kangaroo care) (Yasova Barbeau et al., 2019). Measurements of "body temperature (°C), peak heart rate (min), respiratory rate (min), oxygen saturation (mmHg), blood pressure (mmHg)" of infants and mothers before and after the intervention will be recorded in this chart. The chart was sent to 5 academicians who are experts in Pediatric Nursing and their expert opinions were taken and the chart was finalized by making the necessary changes in line with their suggestions.

OTHER OUTCOMES:
Spielberg State Anxiety Scale | Before starting the study and after completion of the study at the end of 3 days
  The State Anxiety Inventory, which was adapted to Turkish culture by Öner and Le Compte (1983) and norm studies were conducted along with validity and reliability studies, consists of a total of twenty items. The State Anxiety Inventory requires individuals to describe how they feel at a certain moment under certain conditions and to answer the items by taking into account their feelings about the situation they are in. The feelings or behaviors expressed in the items of the State Anxiety Scale are answered by marking one of the options such as (1) not at all, (2) a little, (3) a lot, (4) completely, according to the degree to which the individual feels the situation. Scoring: The scales have "direct (straight)" and inverted expressions. When scoring inverted statements expressing positive emotions, those with a weight value of 1 are converted to 4 and those with a weight value of 4 are converted to 1.

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared upon reasonable request from qualified researchers. Requests will be evaluated by the study investigators, and data will be shared in compliance with ethical and institutional regulations.

REFERENCES:
- [Result] Yasova Barbeau D, Krueger C, Huene M, Copenhaver N, Bennett J, Weaver M, Weiss MD. Heart rate variability and inflammatory markers in neonates with hypoxic-ischemic encephalopathy. Physiol Rep. 2019 Aug;7(15):e14110. doi: 10.14814/phy2.14110. PMID 31397094
- [Result] Öner N, Le Compte A. Durumluk Sürekli Kaygı Envanteri El Kitabı, İstanbul, Boğaziçi Üniversitesi Yayınları, İstanbul, 1983.
- [Result] Butcher NJ, Monsour A, Mew EJ, Chan AW, Moher D, Mayo-Wilson E, Terwee CB, Chee-A-Tow A, Baba A, Gavin F, Grimshaw JM, Kelly LE, Saeed L, Thabane L, Askie L, Smith M, Farid-Kapadia M, Williamson PR, Szatmari P, Tugwell P, Golub RM, Monga S, Vohra S, Marlin S, Ungar WJ, Offringa M. Guidelines for Reporting Outcomes in Trial Reports: The CONSORT-Outcomes 2022 Extension. JAMA. 2022 Dec 13;328(22):2252-2264. doi: 10.1001/jama.2022.21022. PMID 36511921
- [Result] Arnon S, Diamant C, Bauer S, Regev R, Sirota G, Litmanovitz I. Maternal singing during kangaroo care led to autonomic stability in preterm infants and reduced maternal anxiety. Acta Paediatr. 2014 Oct;103(10):1039-44. doi: 10.1111/apa.12744. Epub 2014 Aug 11. PMID 25039678